CLINICAL TRIAL: NCT03001401
Title: Comparison of Next Generation Laser Techniques of Myopia Correction: iDesign vs. SMILE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Narayana Nethralaya (Other)
Responsible Party: Principal Investigator, Dr Rohit Shetty, Doctor, Narayana Nethralaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C/2016/09/07
Record Dates: First submitted 2016-12-15; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iDesign (Active Comparator): Eyes will under LASIK using iDesign platform for treatment of sphere and cylinder power
  Interventions: Other: iDesign
- SMILE (Active Comparator): Eyes will under SMILE using Visumax platform for treatment of sphere and cylinder power
  Interventions: Other: SMILE

INTERVENTIONS:
Other: iDesign — One group will under go standard LASIK using iDesign platform (J&J, USA). Visual acuity, tomography outcomes, biomechanical outcomes and inflammation in myopic eyes treated with iDesign and SMILE are proposed to be evaluated under the study.
  Arms: iDesign
Other: SMILE — The other group will undergo SMILE for treatment refractive error (Carl Zeiss, Germany). isual acuity, tomography outcomes, biomechanical outcomes and inflammation in myopic eyes treated with iDesign and SMILE are proposed to be evaluated under the study.
  Arms: SMILE

SUMMARY:
The proposed study seeks to compare visual acuity, tomographic outcomes, biomechanical changes and inflammatory profile of normal eyes (matched for age, refraction and corneal thickness) undergoing iDesign and SMILE procedure. The hypothesis is that iDesign may deliver equivalent or better clinical outcomes than SMILE, by removing less tissue and correcting for higher order aberrations.

DETAILED DESCRIPTION:
iDesign is a promising new technique to treat myopia with astigmatism using ocular aberrations measured with a high resolution wavefront sensor.[1,2] Early studies with iDesign platform has established its safety and efficacy in correction of myopia with fewer patients reporting night vision problems.[1,2] In keratoconus, iDesign has also provided excellent outcomes following collagen crosslinking.3 SMILE is a recent technique that eliminates creation of flap and appears to achieve similar refractive outcomes as conventional LASIK but with less dryness, less inflammation and faster wound healing.[4,5] SMILE corrects lower order aberrations only.[4,5] Thus, a comparative assessment of iDesign and SMILE is necessary since iDesign can potentially give better visual outcomes with lower volume of tissue removal. If lower volume of tissue is removed, it is also hypothesized that the corneal would be more stable biomechanically.[5] Further, SMILE does not provide any correction of higher order aberrations. With the inclusion of higher order aberrations in the iDesign treatment plan, it is hypothesized that both short and long term outcomes will be better with iDesign than with SMILE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be between 18 to 50 years of age.
2. Patient must have stable myopia for a minimum period of one year (a change of 0.25D or less) as documented by prior clinical records or current spectacle correction.
3. Patient must have a corrected distance visual acuity (CDVA) of 20/25 or better,
4. Patient must have a spherical equivalent refraction less than -10D
5. Patient must have refractive astigmatism less than 3D.

Exclusion Criteria:

1. Patient must not have a central corneal thickness (CCT) less than 480 micrometer
2. Patient must not have a calculated residual stromal bed thickness of less than 250 micrometer after the surgery
3. Patient must not have symptoms or signs of keratoconus, diabetes, collagen vascular disease, pregnancy, breastfeeding and any prior ocular surgery.
4. Patient must not have an inter-ocular difference of more than 1.00 diopter (D) of spherical or 0.50 D of cylindrical refractive error.
5. Patient must not be on chronic systemic steroids or other medication that can affect wound healing.
6. Patient must not be allergic to primary or alternative medications.
7. Patient must not be using rigid contact lenses for the last three weeks or soft contact lenses for at least 1 week before the preoperative evaluation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity measured as Logarithm of manifest refraction | Post surgery over a period of 1 year
  Uncorrected and corrected distance visual acuity

SECONDARY OUTCOMES:
Change in Corneal curvature in Diopter | Post surgery over a period of 1 year
  Optical coherence tomography and Scheimpflug imaging of the cornea will be performed
Change in deformation of the cornea | Post surgery over a period of 1 year
  Air-puff applanation of the cornea will be used to asses deformation
Change in ocular surface dryness and/or pain | Post surgery over a period of 1 year
  Assessed by ocular surface discomfort score
Change in wavefront aberrations described by Zernike Polynomials | Post surgery over a period of 1 year
  Corneal and ocular aberrations

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Shetty, MD, PHD, Principal Investigator — Narayana Nethralaya
Locations (1):
- Narayana Nethralaya, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schallhorn SC, Venter JA, Hannan SJ, Hettinger KA. Outcomes of wavefront-guided laser in situ keratomileusis using a new-generation Hartmann-Shack aberrometer in patients with high myopia. J Cataract Refract Surg. 2015 Sep;41(9):1810-9. doi: 10.1016/j.jcrs.2015.10.007. PMID 26603388
- [Background] Schallhorn SC, Venter JA, Hannan SJ, Hettinger KA. Wavefront-Guided Photorefractive Keratectomy with the Use of a New Hartmann-Shack Aberrometer in Patients with Myopia and Compound Myopic Astigmatism. J Ophthalmol. 2015;2015:514837. doi: 10.1155/2015/514837. Epub 2015 Oct 4. PMID 26504595
- [Background] Shaheen MS, Shalaby Bardan A, Pinero DP, Ezzeldin H, El-Kateb M, Helaly H, Khalifa MA. Wave Front-Guided Photorefractive Keratectomy Using a High-Resolution Aberrometer After Corneal Collagen Cross-Linking in Keratoconus. Cornea. 2016 Jul;35(7):946-53. doi: 10.1097/ICO.0000000000000888. PMID 27191671
- [Background] Denoyer A, Landman E, Trinh L, Faure JF, Auclin F, Baudouin C. Dry eye disease after refractive surgery: comparative outcomes of small incision lenticule extraction versus LASIK. Ophthalmology. 2015 Apr;122(4):669-76. doi: 10.1016/j.ophtha.2014.10.004. Epub 2014 Nov 22. PMID 25458707
- [Background] Reinstein DZ, Archer TJ, Gobbe M. Small incision lenticule extraction (SMILE) history, fundamentals of a new refractive surgery technique and clinical outcomes. Eye Vis (Lond). 2014 Oct 16;1:3. doi: 10.1186/s40662-014-0003-1. eCollection 2014. PMID 26605350
- [Background] McNabb RP, Farsiu S, Stinnett SS, Izatt JA, Kuo AN. Optical coherence tomography accurately measures corneal power change from laser refractive surgery. Ophthalmology. 2015 Apr;122(4):677-86. doi: 10.1016/j.ophtha.2014.10.003. Epub 2014 Dec 6. PMID 25487424
- [Background] Matalia J, Francis M, Tejwani S, Dudeja G, Rajappa N, Sinha Roy A. Role of Age and Myopia in Simultaneous Assessment of Corneal and Extraocular Tissue Stiffness by Air-Puff Applanation. J Refract Surg. 2016 Jul 1;32(7):486-93. doi: 10.3928/1081597X-20160512-02. PMID 27400081
- [Background] Sinha Roy A, Kurian M, Matalia H, Shetty R. Air-puff associated quantification of non-linear biomechanical properties of the human cornea in vivo. J Mech Behav Biomed Mater. 2015 Aug;48:173-182. doi: 10.1016/j.jmbbm.2015.04.010. Epub 2015 Apr 20. PMID 25955559